CLINICAL TRIAL: NCT00535574
Title: Bexarotene Augmentation of Antipsychotic Treatment for Chronic Schizophrenia: a 6-week, Randomized, Double-blind Placebo-controlled Trial
Brief Title: Bexarotene Augmentation of Antipsychotic Treatment for Chronic Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beersheva Mental Health Center (Other Government)
Responsible Party: Principal Investigator, Vladimir Lerner, A/Professor, Head of department, Beersheva Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LRM250850
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2011-05

CONDITIONS: Schizophrenia
Keywords: retinoids; bexarotene; schizophrenia; PANSS; Positive and negative symptoms of schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Bexarotene

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bexarotene (Targretin LGD1069) (Placebo Comparator)
  Interventions: Drug: Bexarotene (Targretin LGD1069); Drug: bexarotene
- placebo (Active Comparator)
  Interventions: Drug: Bexarotene (Targretin LGD1069)

INTERVENTIONS:
Drug: Bexarotene (Targretin LGD1069) — 75 mg per day for 6 weeks
Drug: bexarotene — 75 mg/day 6 weeks
  Arms: Bexarotene (Targretin LGD1069)

SUMMARY:
Background: Bexarotene (Targretin) is a synthetic retinoid mainly used for treatment of patients suffer from oncological or dermatological diseases. The present study is based on: evidence that retinoids are involved in neurodevelopment ("the retinoid dysregulation hypothesis"); an assumption that the combined effect of antipsychotic agents and bexarotene will have a beneficial effect on schizophrenia patients; and the positive findings from our pilot open-label clinical trial (ClinicalTrials.gov Identifier: NCT00141947). However, clinical efficacy of bexarotene should be investigated in a placebo-controlled trial.

Methods: In a 6-week, randomized, double-blind placebo-controlled trial Targretin (75 mg/day) or placebo capsules will be added to the stable ongoing antipsychotic treatment of 90 schizophrenia patients. Participants will be assessed at baseline and after 2, 4 and 6 weeks of treatment. A battery of research instruments will be used for assessment of psychopathology, side effects, general functioning and quality of life. In addition, cholesterol and triglyceride levels, liver and thyroid function tests and a blood cell count will be monitored at baseline and during the study

DETAILED DESCRIPTION:
Recruiting was beginning on November 2008

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60 years, male or female
2. DSM-IV criteria for schizophrenia, or schizoaffective disorder.
3. Ability and willingness to sign informed consent for participation in the study
4. Stable blood parameters including adequate hematologic function, defined as WBC ≥ 4.300/μL, absolute neutrophil count ≥3.000/μL (> 50%), and platelet count ≥ 180,000/μL; normal coagulation parameters; bilirubin ≤1.5 times the upper limit of normal (ULN); AST/ALT ≤ 2.5 × ULN; and serum creatinine ≤1.5 mg/dL.
5. Only patients who had a normal baseline fasting triglyceride (FTG) level will be entered into the study; triglycerides may be normalized before study entry with use of an antilipemic agent.

Exclusion Criteria:

1. Lipid abnormalities. Fasting triglyceride normal (normalization with an antilipemic allowed prior to study entry).
2. Leucopenia or neutropenia. Hematopoietic: Hemoglobin at least 12.5 g/dL; WBC< 4300/μL; Absolute neutrophil count < 3000/μL; Platelet count < 155,000/μL
3. Evidence of organic brain damage, mental retardation, alcohol or drug abuse
4. Impairment of renal function
5. Hepatic dysfunction
6. A history of pancreatitis
7. Thyroid axis alterations
8. Suicide attempt in past year.
9. Cataracts.
10. Systemic treatment with more than 15,000 IU of vitamin A daily.
11. Patients with a known hypersensitivity to bexarotene or other components of the product.
12. Pregnant women or a woman who intends to become pregnant.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2008-11; Primary Completion 2010-12 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
PANSS, CDSS, GAF, QLS | every two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Vladimir Lerner, MD, PhD, Principal Investigator — Be'er Sheva Mental Health Center Ben Gurion University of the Negev
Locations (3):
- Israel (3):
  - Be'er Sheva Mental Health Center, Beersheba, Be'er Sheva
  - Abarbanel Mental Health Center, Bat Yam
  - Sha'ar Menashe Mental Health Center,, Hadera

REFERENCES:
- [Derived] Lerner V, Miodownik C, Gibel A, Sirota P, Bush I, Elliot H, Benatov R, Ritsner MS. The retinoid X receptor agonist bexarotene relieves positive symptoms of schizophrenia: a 6-week, randomized, double-blind, placebo-controlled multicenter trial. J Clin Psychiatry. 2013 Dec;74(12):1224-32. doi: 10.4088/JCP.12m08160. PMID 24434091